CLINICAL TRIAL: NCT04137055
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ZSP0678 and the Effect of Food on ZSP0678 Pharmacokinetics in Chinese Healthy Subjects.
Brief Title: Study in Chinese Healthy Adults to Evaluate the Safety, Tolerability and Pharmacokinetics on ZSP0678, and the Effect of Food on ZSP0678 Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZSP0678-19-01
Record Dates: First submitted 2019-10-15; First posted 2019-10-23 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Nonalcoholic Steatohepatitis
Keywords: NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- ZSP0678-10mg (single dose)-Cohort 1 (Experimental): ZSP0678/Placebo 10mg
  Interventions: Drug: ZSP0678-10mg; Drug: ZSP0678 Placebo
- ZSP0678-30mg (single dose)-Cohort 2 (Experimental): ZSP0678/Placebo 30 mg Enrollment into Cohort 2 will begin upon assurance of safety for Cohort 1.
  Interventions: Drug: ZSP0678-30mg; Drug: ZSP0678 Placebo
- ZSP0678-60mg (single dose)-Cohort 3 (Experimental): ZSP0678/Placebo 60mg Enrollment into Cohort 3 will begin upon assurance of safety for Cohort 2.
  Interventions: Drug: ZSP0678-60mg; Drug: ZSP0678 Placebo
- ZSP0678-120mg (single dose)-Cohort 4 (Experimental): ZSP0678/Placebo 120mg Enrollment into Cohort 4 will begin upon assurance of safety for Cohort 3.
  Interventions: Drug: ZSP0678-120mg; Drug: ZSP0678 Placebo
- ZSP0678-180mg (single dose)-Cohort 5 (Experimental): ZSP0678/Placebo 180mg Enrollment into Cohort 5 will begin upon assurance of safety for Cohort 4.
  Interventions: Drug: ZSP0678-180mg; Drug: ZSP0678 Placebo
- ZSP0678-240mg (single dose)-Cohort 6 (Experimental): ZSP0678/Placebo 240mg Enrollment into Cohort 6 will begin upon assurance of safety for Cohort 5.
  Interventions: Drug: ZSP0678-240mg; Drug: ZSP0678 Placebo
- ZSP0678-320mg (single dose)-Cohort 7 (Experimental): ZSP0678/Placebo 320mg Enrollment into Cohort 7 will begin upon assurance of safety for Cohort 6.
  Interventions: Drug: ZSP0678-320mg; Drug: ZSP0678 Placebo
- ZSP0678 (food effect)-Cohort FE (Experimental): Period 1: Group A and Group B receive ZSP0678/Placebo under the fasting or fed condition ,respectively on Day1.
  Period 2: Group A and Group B receive ZSP0678/Placebo under the fed or fasting condition ,respectively on Day8.
  Enrollment into Cohort FE will begin upon assurance of safety for Cohort 4.
  Interventions: Drug: ZSP0678; Drug: ZSP0678 Placebo
- ZSP0678 Dose1 (multiple doses)-Cohort 8 (Experimental): ZSP0678/Placebo Dose1 will be administrated according to the results of Cohort 2&3
  Interventions: Drug: ZSP0678-Dose 1; Drug: ZSP0678 Placebo
- ZSP0678 Dose2 (multiple doses)-Cohort 9 (Experimental): ZSP0678/Placebo Dose2 will be administrated according to the results of Cohort 3&4
  Interventions: Drug: ZSP0678-Dose 2; Drug: ZSP0678 Placebo
- ZSP0678 Dose3 (multiple doses)-Cohort 10 (Experimental): ZSP0678/Placebo Dose3 will be administrated according to the results of Cohort 4&5
  Interventions: Drug: ZSP0678-Dose 3; Drug: ZSP0678 Placebo

INTERVENTIONS:
Drug: ZSP0678-10mg — ZSP0678 tablet administered orally under fasted condition
  Arms: ZSP0678-10mg (single dose)-Cohort 1
Drug: ZSP0678-30mg — ZSP0678 tablets administered orally under fasted condition
  Arms: ZSP0678-30mg (single dose)-Cohort 2
Drug: ZSP0678-60mg — ZSP0678 tablets administered orally under fasted condition
  Arms: ZSP0678-60mg (single dose)-Cohort 3
Drug: ZSP0678-120mg — ZSP0678 tablets administered orally under fasted condition
  Arms: ZSP0678-120mg (single dose)-Cohort 4
Drug: ZSP0678-180mg — ZSP0678 tablets administered orally under fasted condition
  Arms: ZSP0678-180mg (single dose)-Cohort 5
Drug: ZSP0678-240mg — ZSP0678 tablets administered orally under fasted condition
  Arms: ZSP0678-240mg (single dose)-Cohort 6
Drug: ZSP0678-320mg — ZSP0678 tablets administered orally under fasted condition
  Arms: ZSP0678-320mg (single dose)-Cohort 7
Drug: ZSP0678 — ZSP0678 tablets administered orally under fasted or fed condition
  Arms: ZSP0678 (food effect)-Cohort FE
Drug: ZSP0678-Dose 1 — ZSP0678 tablets administered orally once daily for 14 Days
  Arms: ZSP0678 Dose1 (multiple doses)-Cohort 8
Drug: ZSP0678-Dose 2 — ZSP0678 tablets administered orally once daily for 14 Days
  Arms: ZSP0678 Dose2 (multiple doses)-Cohort 9
Drug: ZSP0678-Dose 3 — ZSP0678 tablets administered orally once daily for 14 Days
  Arms: ZSP0678 Dose3 (multiple doses)-Cohort 10
Drug: ZSP0678 Placebo — Participants will receive placebo matching to ZSP0678 orally.

SUMMARY:
This study will evaluate the safety, tolerability and pharmacokinetics (PK) of escalating single-and multiple-oral doses of ZSP0678 on fasted condition, and characterize PK of ZSP0678 on an empty stomach (fasted condition) and following a high fat, high calorie meal (fed condition) in a 2-period, 2-sequence manner. The study will be conducted in 3 parts (Ascending single dose, multiple dose and food effect). Participants will receive either ZSP0678 or placebo .

ELIGIBILITY:
Inclusion Criteria:

* Subjects are required to meet the following criteria in order to be included in the trial:

  1. Signature signed informed consent before the trial, and fully understood the content, process and possible adverse reactions.
  2. Subjects must be willing and able to complete the research according to the experimental protocol.
  3. Subjects (including partners) are willing to take effective contraceptive measures and have no pregnancy plan during the whole study period until 6 months after drug withdrawal.
  4. Male and female subjects aged 18-50 (including 18 and 50)
  5. Body weight of male subjects should not be less than 50kg and that of female subjects should not be less than 45kg.Body mass index (BMI) = weight (kg)/height 2 (m2), the range of 19~26kg/m2 (including the critical value);
  6. Physical condition:No significant abnormalities in medical history, including cardiovascular system, liver, kidneys, gastrointestinal system, neural system, respiratory system (eg.asthma,asthma induced by exercise,chronic obstructive pulmonary disease), mental, metabolism, etc.
  7. Subjects in general good health or No significant abnormalities in the opinion of the investigator as determined by vital signs and a physical examination.

     Exclusion Criteria:
* Eligible subjects must not meet any of the following exclusion criteria:

  1. Allergic constitution (allergic to many drugs, especially to ingredients similar to the test drug and food)
  2. The average daily smoking are more than 5 cigarettes within 3 months prior to screening.
  3. Known history of drug or alcohol abuse.(defined as consumption of more than 30g of ethanol a day for male and more than 20 g for female )
  4. Subjects who donated blood or bleeding profusely(> 400 mL)in the 3 months preceding study screening.
  5. History of dysphagia or any gastrointestinal illness that affects drug absorption, including a history of frequent nausea or vomiting from any cause, irregular gastrointestinal motility, such as habitual diarrhea, constipation, or irritable bowel syndrome.
  6. History or presence of any disease or condition known to increase the risk of bleeding, eg.acute gastritis, duodenal ulcer, etc.
  7. Participated in another clinical research study and received any investigational products within 3 months prior to dosing.
  8. Use of any prescription or over-the-counter (OTC) medications, vitamins and herbal within 14 days prior to screening.
  9. History of having any special food(including dragon fruit, mango, grapefruit, etc.),strenuous exercises,or other factors may interfere with the absorption, distribution, metabolism, or excretion of drug within 14 days prior to screening.
  10. Subjects who cannot tolerate standard meals (this clause only applies to subjects participating in food impact studies).
  11. Presence of clinically significant abnormalities in ECG or QTcB>450ms in males,or QTcB>470ms in females.
  12. Pregnancy or breastfeeding at screening and during the study.All female subjects of childbearing potential must have a negative urine pregnancy test at screening and during the trial.
  13. Any clinically significant abnormality upon physical examination or in the clinical laboratory tests. History or presence of a clinically significant gastrointestinal, renal, hepatic, neurologic, hematic, endocrine, neoplastic, pulmonary, immune, psychiatric or cardiovascular and cerebrovascular disorder(s) (but not limited to above disorders).
  14. Presence of human immunodeficiency virus (HIV), viral hepatitis(including hepatitis C virus (HCV) or hepatitis B virus (HBV) ),treponema pallidum antibodies at screening.
  15. Any acute illness or concomitant medication from screening to first dosing.
  16. Have chocolate, any food or beverage that contains caffeine ,xanthine and alcohol within 24 hours prior to dosing.
  17. Positive for urine drug screening or history of substance abuse for a period of 5 consecutive years before screening.
  18. As judged by the researcher, it is not suitable to join the clinical researcher.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Number and severity of adverse events (AEs) and Serious Adverse Events(SAE) following oral doses of ZSP0678 and placebo. | SAD Group: Up to 5 days, MAD: Up to 18 days, FE group: Up to11 days after first dose ]
Tmax | UP to 5, 18, 11 days for SAD, MAD, FE part respectively
  The time after dosing when Cmax occurs
Cmax | UP to 5, 18, 11 days for SAD, MAD, FE part respectively
  Maximum concentration
t1/2 | UP to 5, 18, 11 days for SAD, MAD, FE part respectively
  t1/2 is defined as the time to decline half of the drug concentration in plasma.
AUCinf（AUC0-∞） | UP to 5, 18, 11 days for SAD, MAD, FE part respectively
  Area under the curve extrapolated until time is infinity (AUCinf)
AUClast（AUC0-t） | UP to 5, 18, 11 days for SAD, MAD, FE part respectively
  AUClast is defined as the concentration of drug from time zero to the last quantifiable concentration.
CL/F | UP to 5, 18, 11 days for SAD, MAD, FE part respectively
  CL/F is defined as the ratio of total clearance(Cl) to bioavailability(F).
λz | UP to 5, 18, 11 days for SAD, MAD, FE part respectively
  λz is defined as the ratio between the elimination of compound per unit time and the total amount of compound.
CLr | UP to 5, 18, 11 days for SAD, MAD, FE part respectively
  CLr is defined as how many milliliters of plasma in which some substance can be completely eliminated in the unit time (per minute) of two kidneys.
Multiple-dose plasma PK parameter: Rac of ZSP0678 at steady state | UP to 18 days.
  Rac (Accumulation Index) is defined as the ratio between AUC0-XX in Day XX and AUC0-XX in Day1
Multiple-dose plasma PK parameter: DF of ZSP0678 at steady state | UP to 18 days.
  DF is defined as the percentage of fluctuation in steady state is 100 * (Cmax, ss - Cmin, ss)/Cavg, ss.
Multiple-dose plasma PK parameter: Cmin of ZSP0678 at steady state | UP to 18 days.
  Cmin is defined as the minimum observed concentration of drug in plasma at steady state.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital Affiliated to Capital Medical Universit, Beijing, Beijing Municipality, China